CLINICAL TRIAL: NCT02873819
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Determine the Safety and Efficacy of GL-0817 (With Cyclophosphamide) for the Prevention of Recurrence in HLA-A2+ Patients With High-Risk Squamous Cell Carcinoma of the Oral Cavity
Brief Title: Safety and Efficacy Study of GL-0817 (With Cyclophosphamide) for the Prevention of Recurrence of Squamous Cell Carcinoma of the Oral Cavity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gliknik Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GL0817-01; 2016-001256-22 (EudraCT Number)
Record Dates: First submitted 2016-08-08; First posted 2016-08-22 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2020-09

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — poly ICLC; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GL-0817 (Experimental): Subjects in active treatment will be vaccinated with GL-0817 with the adjuvants Poly-ICLC (Hiltonol®) and GM-CSF (Sargramostim, Leukine®) 3 times at 3-week intervals followed by 7 doses at 3-month intervals beginning at Week 18. Patients will receive IV Cyclophosphamide 1 day prior to the first 3 vaccinations.
  Interventions: Drug: GL-0817; Drug: Hiltonol; Drug: Sargramostim; Drug: cyclophosphamide
- Placebo (Placebo Comparator): Subjects in placebo arm will receive placebo to cyclophosphamide (normal saline solution) followed by Poly-ICLC/GM-CSF/placebo vaccine injections on the same schedule as the GL-0817 cohort.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GL-0817 — GL-0817, IV at the dose 1.5 mg will be administered 3 times at 3-week intervals followed by 7 doses at 3-month intervals beginning at the Week 18 visit
  Other Names: Biropepimut-S
  Arms: GL-0817
Drug: Hiltonol — Hiltonol will be administered intramuscularly at the dose of 1.4 mg as adjuvant to GL0817, 3 times at 3-week intervals followed by 7 doses at 3-month intervals beginning at the Week 18 visit
  Other Names: Poly-ICLC
  Arms: GL-0817
Drug: Sargramostim — Sargramostim will be administered intramuscularly at the dose of 100 μg/m2, as adjuvant to GL0817, 3 times at 3-week intervals followed by 7 doses at 3-month intervals beginning at the Week 18 visit
  Other Names: GM-CSF; Leukine
  Arms: GL-0817
Drug: cyclophosphamide — cyclophosphamide will be administered IV at a dose of 200 mg/m2 (maximum dose 400 mg) one day prior to first three vaccinations of GL0817 with adjuvants
  Arms: GL-0817
Drug: Placebo — Placebo (normal saline) will be administered as per the schedule of cyclophosphamide and GL0817/adjuvants administration
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind clinical trial to assess the safety and efficacy of GL-0817 as a means to prevent disease recurrence in patients considered at high-risk following surgery and adjuvant chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Histologic diagnosis of squamous cell carcinoma of the oral cavity including the lip, floor of mouth, anterior 2/3 of tongue, alveolus and gingiva, buccal mucosa, hard palate and retromolar trigone
3. Subjects must have undergone primary gross total resection (no re-resected patients are allowed) with fulfillment of at least 1 of the following histologic criteria for high-risk disease:

   * Histologic involvement of 2 or more regional lymph nodes
   * Any lymph node with histologic extracapsular extension (ECS)
   * Close (<3mm) or positive surgical margins on microscopic evaluation with no gross residual tumor
4. No evidence of locoregional disease or distant metastases at screening. Subjects must have negative scans (CT, CT-PET or MRI) for locoregional recurrence, brain or lung metastases. A negative biopsy will be mandated in patients with a positive scan. Other evaluations should be performed as clinically indicated.
5. No history of distant metastases.
6. Tumor tissue from surgery or biopsy must be available to determine MAGE-A3 expression for correlative studies.
7. Following surgery, the patient must have received external beam radiotherapy (58-66 Gy in 2 Gy fractions, 5 days per week) with concomitant cisplatin starting within 8 weeks of surgery. A brief delay in the initiation of radiotherapy following 8 weeks post-surgery due to administrative reasons (e.g., start of RT on Mondays) may be permitted by the Medical Monitor. The cumulative dose of cisplatin the subject received must be > 150 mg/m2. Protocol therapy must be initiated within a period of 4-8 weeks (28-56 days) following the end of RT.
8. The patient is, in the investigator's opinion, adequately recovered from the effects of surgery and chemoradiotherapy to participate in this study.
9. Blood HLA-A2 phenotype
10. ECOG Performance Status < 1
11. Laboratory values obtained ≤ 14 days prior to randomization:

    * Absolute neutrophil count (ANC) ≥ 1500/μL (without intervention, e.g., G-CSF)
    * Platelets ≥ 75,000/μL (without intervention, e.g., transfusion)
    * Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥8.0 g/dl is acceptable).
    * Alkaline phosphatase ≤ 2.5 x upper limit of normal (ULN)
    * AST and ALT ≤ 2 x ULN
    * Creatinine < 2 x ULN
    * Bilirubin < 1.5x ULN (except for patients with Gilbert's disease, for whom the upper acceptable limit of serum bilirubin is 3mg/dL)
12. A female subject is eligible to enter the study if she is:

    * not pregnant or nursing; Female participants must not breastfeed during the study and for a period of 30 days following the last dose.
    * of non-childbearing potential (i.e., women who had a hysterectomy, are postmenopausal which is defined as 1 year without menses, have both ovaries surgically removed or have current documented tubal ligation); or
    * of childbearing potential (i.e., women with functional ovaries and no documented impairment of oviductal or uterine function that would cause sterility). This category includes women with oligomenorrhea [even severe], women who are perimenopausal or have just begun to menstruate. These women must have a negative serum pregnancy test at screening, and agree to one of the following:

      * complete abstinence from intercourse from 2 weeks prior to administration of the 1st dose of study agent and 6 months after the last dose of study agent; or
      * consistent and correct use of 1 of the following highly effective methods of birth control for one month prior to the start of the study agent and 6 months after the last dose:
    * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
    * progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
    * intrauterine device (IUD)
    * intrauterine hormone-releasing system ( IUS)
    * bilateral tubal occlusion
    * vasectomized partner (if vasectomized is the sole sexual partner and has received medical confirmation of surgical success)
13. A male subject who is sexually active with a woman of childbearing potential is eligible to enter the study if he agrees to use effective contraception throughout the study and for 6 months after the last dose of study agent.
14. The subject must be capable of understanding the investigational nature, potential risks and benefits of the study and capable of providing valid informed consent. The subject must provide study specific informed consent prior to any protocol procedures that are not a part of standard care, including consent for assessment of HLA-A2 status, mandatory tissue submission for MAGE-A3 analysis and correlative studies.
15. The subject must be willing to return to the study center for vaccinations and study-related follow up procedures including blood and tumor collections and completion of imaging studies as required by the protocol.

Exclusion Criteria:

1. Known HIV or hepatitis B/C infection (testing not required). Subjects who are hepatitis C antibody positive may be enrolled if they are confirmed to have a negative viral load at screening.
2. Subjects with active autoimmune disease or a history of autoimmune disease requiring systemic steroids or other immunosuppressive treatment.
3. Subjects who have used systemic corticosteroids or other immunosuppressants for any condition within 14 days of randomization. Inhaled or topical steroids are permitted.
4. Any medical condition which would, in the investigator's opinion, compromise the patient's ability to mount an immune response, renders the patient a poor candidate for this trial or could confound the results of the study
5. Major surgery or traumatic injury within 28 days of randomization
6. Prior splenectomy or organ allograft
7. Any other prior, concurrent or planned chemotherapy, immunotherapy, radiotherapy, device, or investigational therapy for this cancer other than those specified in this study.
8. History of other malignancy (i.e., excluding disease under study) within 3 years of randomization. Exceptions include: adequately-treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix or breast, or adequately treated non-metastatic prostate cancer.
9. Known hypersensitivity to GM-CSF, yeast-derived products or any component of the GM-CSF drug product (e.g., mannitol) or poly-ICLC (e.g., carboxymethylcellulose).
10. Known hypersensitivity to cyclophosphamide, its metabolites or any other components, or known urinary outflow obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Disease-free interval | Up to 2 years

SECONDARY OUTCOMES:
Disease-free survival (DFS) | up to 2 years
Overall survival (OS) | up to 5 years
Disease-free interval in a per protocol analysis | up to 2 years
Adverse event profile | up to week 94

CONTACTS AND LOCATIONS:
Locations (33):
- University of Maryland Greenebaum Cancer Center, Baltimore, Maryland, United States
- Hungary (5):
  - National Institute of Oncology, Budapest
  - Semmelweis University, Budapest
  - University of Debrecen Clinical Center, Debrecen
  - Bacs-Kiskun County Teaching Hospital, Kecskemét
  - Medical Center of the University of Pecs, Pécs
- Poland (2):
  - Oncology Center of Prof. Franciszek Lukaszczyk in Bydgoszcz, Bydgoszcz
  - Swietokrzyskie Oncology Center in Kielce, Kielce
- Russia (8):
  - Clinical Oncology Center, Omsk
  - Rostov Oncology Research Institute, Rostov-on-Don
  - Leningrad Regional Oncology Center, Saint Petersburg
  - Oncology Center of Moskovskiy District, Saint Petersburg
  - Ogarev Mordovia State University, Saransk
  - Clinical Hospital #1, Sterlitamak
  - Republican Clinical Oncology Center, Ufa
  - Regional Clinical Oncology Hospital, Yaroslavl
- Serbia (3):
  - Institute of Oncology and Radiology of Serbia, Belgrade
  - Military Medical Academy, Clinic of Maxillofacial Surgery, Belgrade
  - Oncology Institute of Vojvodina (IOV), Clinic of Medical Oncology, Kamenitz
- Spain (3):
  - University Hospital Vall d'Hebron (HUVH), Barcelona
  - University Hospital La Paz, Madrid
  - Parc Tauli Health Corporation, Sabadell
- Ukraine (11):
  - Cherkasy Regional Oncology Center, Cherkasy
  - Chernihiv Regional Oncology Center, Chernihiv
  - Dnipropetrovsk I.I. Mechnykov Regional Clinical Hospital, Dnipro
  - Ivano-Frankivsk Regional Oncology Center, Ivano-Frankivsk
  - Communal Non-profit enterprise "Regional Center of Oncology", Kharkiv
  - Kyiv Regional Oncology Center, Kyiv
  - Lviv Regional Clinical Hospital, Lviv
  - Odesa Regional Oncology Center, Odesa
  - Poltava Regional Clinical Oncology Center, Poltava
  - Sumy Regional Clinical Oncology Center, Sumy
  - Podillia Regional Oncology Center, Vinnytsia

IPD SHARING:
Plan to Share IPD: No